CLINICAL TRIAL: NCT05390632
Title: Head-to-head Comparison Between [18F]-FDG PET/CT and PET/MRI in Lymphomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Xuejuan Wang, Principal Investigator, Peking University Cancer Hospital & Institute
Other Study IDs: XW-PET/CT &PET/MRI-001
Record Dates: First submitted 2022-05-22; First posted 2022-05-25 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: PET/MRI
Keywords: Positron-Emission Tomography; lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigating the performance of 18F-FDG PET/CT and PET/MRI in lymphomas

DETAILED DESCRIPTION:
In this study investigators evaluated Nodal and Extranodal Lymphoma Lesions uptake by 18F-FDG PET (PET/CT and PET/MR). Prior to treatment, all patients will undergo whole-body 18F-FDG PET/CT and PET/MR. The methods' efficiency was compared in the diagnosis of lymph node (LN) and organ involvement.

ELIGIBILITY:
Inclusion Criteria:

* pathologically diagnosed as lymphoma; Written informed consent for receiving PET/MRI after PET/CT examinations. cancer planned chemotherapy or immunotherapy scheme. expected survival ≥ 12 weeks

Exclusion Criteria:

* cannot lie supine for half an hour; refuse to join the clinical researcher; severe liver or kidney dysfunction pregnancy or lactation

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients pathologically diagnosed as lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
SUVmax | 150 days
  Standardized uptake value of 18F-FDG PET/CT and PET/MRI for target lesion of subject or suspected tumor in each time point window (SUV)

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Yang, PhD, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Card Holder's Billing State / Province, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Yuan T, Wei M, Yu B, Zhou N, Zhu H, Yang Z, Wang X. Diagnostic performance of integrated whole-body 18F-FDG PET/MRI for detecting bone marrow involvement in indolent lymphoma: Comparison with 18F-FDG PET or MRI alone. Front Oncol. 2023 Mar 13;13:1136687. doi: 10.3389/fonc.2023.1136687. eCollection 2023. PMID 36994205